CLINICAL TRIAL: NCT01772498
Title: Heart Rate Variability Biofeedback for Psychologically Distressed Brain Tumour Survivors
Brief Title: HRV Biofeedback for Brain Tumour Survivors
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRVB-123
Record Dates: First submitted 2012-12-04; First posted 2013-01-21 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Depression; Anxiety; Sleep Impairment
Keywords: depression; anxiety; sleep; pain; biofeedback; breathing; resonant
MeSH Terms: conditions — Depression; Anxiety Disorders; Pain; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heart rate variability biofeedback (Experimental): Heart rate variability biofeedback training administered in eight, individual, weekly, one hour sessions. There will also be 20 minutes a day of resonant frequency breathing to be conducted at home. This intervention involves teaching subjects how to breath at their resonant frequency in a relaxed, diaphramatic manner.
  Interventions: Behavioral: heart rate variability biofeedback

INTERVENTIONS:
Behavioral: heart rate variability biofeedback
  Other Names: resonant frequency biofeedback; RSA biofeedback

SUMMARY:
This study is designed to take a first step toward testing the efficacy and acceptability of heart rate variability biofeedback (HRVB) as a means of ameliorating psychological distress in survivors of Primary Brain Tumour (PBT). HRVB is a biofeedback approach that provides clients with real time feedback about their heart rate variability (HRV) as a means of teaching them how to breathe in a specific, therapeutic manner.

More specifically, this study has been designed to test several hypothesises. Each hypothesis is based on the prediction that, in a sample of psychologically distressed PBT survivors, a course of 8 HRVB sessions will demonstrate:

* statistically significant reductions in levels of depression
* statistically significant reductions in levels of anxiety
* statistically significant increases in resting HRV
* that reductions in anxiety and depression will be significantly, negatively correlated with increases in resting HRV
* that the HRVB will be viewed as an acceptable intervention by the participants

In addition to the hypothesises stated above, the study will also investigate in a discovery oriented manner if the HRVB intervention will have positive impacts on the participants:

* levels of sleep impairment
* levels of pain

DETAILED DESCRIPTION:
Purpose

This study will test the efficacy and acceptability of heart rate variability biofeedback (HRVB) as a means of ameliorating psychological distress in survivors of Primary Brain Tumour (PBT). HRVB is a biofeedback approach that provides clients with real time feedback about their heart rate variability (HRV) as a means of teaching them how to breathe in a specific, therapeutic manner. HRVB has been shown to increase autonomic nervous system efficiency and also to decrease both anxiety and depression.

Background Rationale

Anxiety and depression are two of the strongest drivers of overall quality of life (Q of L) in survivors of primary, malignant brain tumour (PMBT). In a cohort of 73 PMBT survivors, "depression scores alone accounted for more than half of the all variance in Q of L scores" (Pelletier et al, 2003, p. 47). Anxiety symptoms were similarly negatively correlated with over-all Q of L(r = -..72) in brain tumour survivors (Janda et al., 2007). Evidence also suggests that, relative to the general population, brain tumour survivors exhibit much higher rates of both depression (Wellisch et al., 2002)and anxiety (Arnold et al., 2007).

Despite these striking findings around the prevalence and importance of anxiety and depression in the brain tumour population, not a single identified study has used a purely psychological intervention to ameliorate symptoms of depression and/or anxiety in this unique, understandably distressed population. Therefore, research of this kind is urgently needed.

Heart Rate variability Biofeedback

A course of HRVB, or some close variant of it, has shown statistically significant effects on depression and/or anxiety in numerous studies. HRVB has also recently been found to associated with improvements in pain and insomnia, two other common barriers to quality of life in PMBT survivors.

Design

Overview

As a very early stage study, a one group, open label design has been adopted.

Recruitment Process

Participants will be recruited by sending letters to potential participants identified through the BC Cancer Agency registry and by encouraging referrals from local oncologists.

Measures

The primary outcome measures will be resting HRV, the Beck Depression Inventory II, the Trait Anxiety Inventory. Secondary outcome will include the Short Form McGill Pain Questionnaire and the Pittsburgh Sleep Quality Index. Likert scale questionnaires will also be used after the intervention to assess the acceptability of the intervention.

HRVB Protocol

The protocol will involve 8 weekly sessions of up to 60 minutes each, following the general approach described by Lehrer, Vaschillo, & Vaschillo (2000). Participants will also practice breathing at their resonant frequency for 20 minutes each day at home.

Analysis

Three forms of analysis will be conducted. First, paired t-tests of residualized changes scores and effect sizes (Cohen's d) will be used to analyze pre-post changes on all of the psychometric measures and on the HRV data. Second, correlational analysis will also be used to see if there are expected associations between pre-post changes in emotion, pain and sleep measures relative to pre-post changes in resting HRV indices. Finally, means and standard deviations will be used to assess participants' likert ratings on the acceptability of the intervention.

Plans for Current Findings

Results will be developed for publication in relevant, peer reviewed scientific journals. Results will also be used to develop future research in this line, including studying the effciacy of HRVB with psychologically distressed caregivers of PMBT survivors.

ELIGIBILITY:
Inclusion Criteria:

* be a survivor of a primary, malignant brain tumour (WHO grades II-IV)
* not have undergone any major treatment (chemotherapy, radiation, surgery) for previous three months
* be psychologically distressed as indicated by a score of 11 or over on either the anxiety or depression subscale of the Psychosocial Screening Instrument for Cancer (PSSCAN)
* be functionally capable of engaging in a time consuming study of this kind, (as indicated by a Karnofsky Scale score of 70/100)

Exclusion Criteria:

* being incompetent to give consent independently
* being actively suicidal (as per a score of 2 or above on the 1-5 point PSSCAN suicidality measure)
* being actively delusional or psychotic
* being judged, by the PI, to be too acutely distressed to benefit from and/or to successfully complete the intervention (e.g. scoring above 20 on either the depression or anxiety scale of the PSSCAN and/or , in the PI's clinical judgment, being without adequate supports or resources in place to adequately manage their current level of distress successfully enough to benefit from and/or to successfully complete the intervention)
* being currently engaged in psychotherapy or another psychologically based treatment that is specifically designed to ameliorate psychological distress

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-08 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in score on Beck Depression Inventory II at 8 weeks | comparison of scores immediately pre-intervention and then immediately post-intervention (8 weeks later)
  Widely used self report measure to assess for symptoms of depression.
Change from baseline scores on trait form of the State Trait Anxiety Inventory (Spielberger et al., 1983)at 8 weeks | comparison of scores immediately pre-intervention and then immediately post-intervention (8 weeks later)
  The Trait Anxiety Inventory is a widely used self report measure of anxiety symptoms.
Change from baseline in resting HRV High Frequency Power | comparison of scores immediately pre-intervention and then immediately post-intervention (8 weeks later)
  Baseline level of High Frequency HRV power (0.15-0.4 Hz) measured in ms2/Hz recorded over 5 minutes of rest at pre-intervention compared to level of High Frequency HRV power (0.15-0.4 Hz) measured in ms2/Hz recorded over 5 minutes of rest recorded aqt post-intervention
Resting Low Frequency HRV power (0.04-0.15 Hz) | comparison of scores immediately pre-intervention and then immediately post-intervention (8 weeks later)
  Baseline level of Low Frequency HRV power (0.15-0.4 Hz) measured in ms2/Hz recorded over 5 minutes of rest at pre-intervention compared to level of Low Frequency HRV power (0.04-0.15 Hz)measured in ms2/Hz recorded over 5 minutes of rest recorded aqt post-intervention
Change in the standard deviation of all NN intervals from baseline in resting heart beat | comparison of scores immediately pre-intervention and then immediately post-intervention (8 weeks later)
  This metric measures the standard deviation of normal beat-to-beat intervals (SDNN) that are present within the heart rythm. it is a time domain measure of HRV and it serves as a marker of overall adaptability of the nervous system.
Subjective Acceptability ratings | To be completed immediately post-intervention (8 weeks after the intiation of training)
  This will be a 5 point Likert scale asking how acceptable the participants found the experience of particiapting in the intervention to be , from "not at all acceptable" to "very acceptable".

SECONDARY OUTCOMES:
Change from baseline score on the Short Form McGill Pain Questionnaire (SFMPQ)(Melzack, 1987) | comparison of scores immediately pre-intervention and then immediately post-intervention (8 weeks later)
  The SFMPQ is a widely used measure of pain related experience.
Change from baseline in scores on the Pittsburgh Sleep Quality Index (Buysse et al., 1989) | comparison of scores immediately pre-intervention and then immediately post-intervention (8 weeks later)
  The Pittsburgh Sleep Quality Index (Buysse et al., 1989)is a widely used self report measure of sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Linden, PhD, Principal Investigator — UBC Department of Psychology
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Pelletier G, Verhoef MJ, Khatri N, Hagen N. Quality of life in brain tumor patients: the relative contributions of depression, fatigue, emotional distress, and existential issues. J Neurooncol. 2002 Mar;57(1):41-9. doi: 10.1023/a:1015728825642. PMID 12125966
- [Background] Janda M, Steginga S, Langbecker D, Dunn J, Walker D, Eakin E. Quality of life among patients with a brain tumor and their carers. J Psychosom Res. 2007 Dec;63(6):617-23. doi: 10.1016/j.jpsychores.2007.06.018. PMID 18061752
- [Background] Wellisch DK, Kaleita TA, Freeman D, Cloughesy T, Goldman J. Predicting major depression in brain tumor patients. Psychooncology. 2002 May-Jun;11(3):230-8. doi: 10.1002/pon.562. PMID 12112483
- [Background] Arnold SD, Forman LM, Brigidi BD, Carter KE, Schweitzer HA, Quinn HE, Guill AB, Herndon JE 2nd, Raynor RH. Evaluation and characterization of generalized anxiety and depression in patients with primary brain tumors. Neuro Oncol. 2008 Apr;10(2):171-81. doi: 10.1215/15228517-2007-057. Epub 2008 Feb 26. PMID 18314416
- [Background] Lehrer PM, Vaschillo E, Vaschillo B. Resonant frequency biofeedback training to increase cardiac variability: rationale and manual for training. Appl Psychophysiol Biofeedback. 2000 Sep;25(3):177-91. doi: 10.1023/a:1009554825745. PMID 10999236